CLINICAL TRIAL: NCT03606876
Title: A Randomized, Double-blinded, Single-dose, 3-arm Parallel, Comparative Study to Evaluate the Pharmacokinetics and Safety of BAT1806 Injection vs Actemra® in Healthy Chinese Male Subjects
Brief Title: Comparative Study to Evaluate the Pharmacokinetics of BAT1806 vs Actemra® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-1806-001-CR
Record Dates: First submitted 2018-07-12; First posted 2018-07-31 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAT1806 injection (Experimental): BAT1806 injection: 4 mg/kg, intravenous infusion over 60 min
  Interventions: Drug: BAT1806 injection
- Actemra(EU-licensed) (Active Comparator): Actemra(EU-licensed): 4 mg/kg, intravenous infusion over 60 min
  Interventions: Drug: BAT1806 injection
- Actemra(US-licensed) (Active Comparator): Actemra(US-licensed): 4 mg/kg, intravenous infusion over 60 min
  Interventions: Drug: BAT1806 injection

INTERVENTIONS:
Drug: BAT1806 injection — Each subject will receive single intravenous drip of 4 mg/kg BAT1806 Injection or Actemra® (EU-licensed and US-licensed).
  Other Names: Actemra(EU-licensed); Actemra(US-licensed)

SUMMARY:
It is a randomized, double-blinded, single-dose, 3-arm parallel, comparative study to evaluate the pharmacokinetics, safety and immunogenicity of BAT1806 Injection vs Actemra® (EU-licensed and US-licensed) in healthy Chinese male subjects. A total of 138 subjects are planned to be included and randomized at a ratio of 1:1:1 to receive single intravenous drip of 4 mg/kg BAT1806 Injection or Actemra® (EU-licensed and US-licensed).

The study has a screening period of 7 days. PK blood samples will be collected from subjects to determine the serum concentration of tocilizumab, thus to evaluate the change and similarity of the pharmacokinetics of the three study drugs.

The investigator will perform safety evaluation for vital signs, physical examinations, injection site reaction, ECG, clinical laboratory tests and adverse events throughout the study. Immunogenicity evaluation (ADA, ADA titration and nAb) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Inform Consent Form and fully understood the trial conduction, procedure and potential adverse reactions before entering the trial;
* Willing and able to follow the visits, treatments specified in this study;
* Subjects (including their partners) who are willing to refrain from pregnancy, sperm donation and take effective contraceptive method in the future 6 months (i.e. 6 months after study medication), see Appendix 4 for specific contraceptive methods;
* Healthy male subjects at age of 18-55 years (inclusive for both);
* BMI between 18-28 kg/m2 (inclusive for both) and body weight between 55-85 kg (inclusive for both);
* Normal physical examinations results or abnormality without clinical significance.

Exclusion Criteria:

* Daily smoking amount of >5 cigarettes within 3 months prior to the trial;
* Any current or history of severe allergic reaction to foods or drugs and History of allergy to tocilizumab or severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies.
* Having a history of alcoholism (14 units of alcohol per week: 1 unit= 285 mL beer, or 25 mL spirit, or 125 mL wine);
* Having donated blood or loss of massive blood (> 450 mL) within 3 months prior to screening, or planning to donate blood or to receive surgery during the study;
* Prior use of prescription medication, over-the-counter drugs, any vitamin products or herbs within 28 days before screening;
* Having significant changes in diet and exercise habits within 2 weeks before screening or from screening to dose;
* Having any diseases that increase the risk of bleeding, such as hemorrhoids with bleeding symptoms, acute gastritis or gastric and duodenal ulcers;
* Color Doppler echocardiography abnormalities with clinical significance;
* Having clinically significant laboratory abnormalities or other clinically indicated diseases (including but not limited to gastrointestinal, renal, liver, neurological, hematological, endocrine, tumor, lung, immune, mental or cardiovascular diseases);
* Ineligible subjects based on investigator's judgement.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoint | 0-2months
  AUC0-inf

SECONDARY OUTCOMES:
Pharmacokinetics Endpoint | 0-2months
  AUC0-t
Pharmacokinetics Endpoint | 0-2months
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: yanhua ding, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Only one site study

REFERENCES:
- [Derived] Ebbers HC, Taylor PC, Leng X, Wei W, Kinsella NM, Zhou Y, Yang X, Chamberlain P. A Comparison of the Immunogenicity of Intravenous BAT1806, a Tocilizumab Biosimilar, and Its Reference Product. Rheumatol Ther. 2025 Jun;12(3):529-546. doi: 10.1007/s40744-025-00760-y. Epub 2025 Apr 8. PMID 40198544
- [Derived] Zhang H, Wang H, Wei H, Chen H, Liu J, Li C, Zhu X, Li X, Yu J, Zhou Y, Yang X, Wang Z, Wu M, Ding Y. A Phase I Clinical Study Comparing the Tolerance, Immunogenicity, and Pharmacokinetics of Proposed Biosimilar BAT1806 and Reference Tocilizumab in Healthy Chinese Men. Front Pharmacol. 2021 Jan 25;11:609522. doi: 10.3389/fphar.2020.609522. eCollection 2020. PMID 33569002